CLINICAL TRIAL: NCT03888885
Title: Effect of Sport Education Intervention in University Required Physical Education: Cluster Randomized Trial of Students' Perceived Physical Literacy and Physical Activity Levels
Brief Title: Effect of Sport Education in University Required PE on Students' Perceived Physical Literacy and Physical Activity Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Choi Siu Ming, PhD Student, Department of Sports Science and Physical Education, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSMing
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Results first posted 2022-07-05 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Physical Activity; Motivation
Keywords: Physical Education; Sport Education; Physical Literacy; Physical Activity; University Students
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sport Education Group (Experimental): Participants participated in the required physical education lessons which were delivered in a season of sport education model for 10 lessons.
  Interventions: Behavioral: Sport Education Model
- Control Group (No Intervention): Participants received no intervention treatment. They were asked to attend in normal physical education classes for the same period of time.

INTERVENTIONS:
Behavioral: Sport Education Model — A total number of 25 lecturers participated in the 12-hour CPD workshop on Sport Education curriculum on June 2018. The content of the workshop focused on the development of a Sport Education season, the changing roles of teachers and students, the assessment of personal and social responsibility, and the application of sport education season and related pedagogies on handball, badminton, swimming and physical conditioning. The Sport Education courseware and class materials were then designed by the eligible lecturers. The intervention was lasted for 10-lesson, 1-day per week and the duration for each lesson was around 90 minutes. The specific five phases in Sport Education model of team selection, teacher-directed, pre-season, formal competition and cumulating event were included. The eligible lecturers led the lessons according to the designated course wares and lesson plans for each sport.
  Arms: Sport Education Group

SUMMARY:
This project examines the effects of implementing sport education model in university required physical education lessons on perceived physical literacy and physical activity levels of the students.

DETAILED DESCRIPTION:
Scholars suggested the practical application of sport education could operationalize physical literacy that some features of this pedagogical model are positively associated to the development and attributes of physical literacy. However, there is no further supplement on the curriculum and pedagogical method for physical educators to develop students as physically literate individuals. Compared to primary school students and adolescents, university students are at the stage of transition from compulsory physical education in secondary school to more self-initiated physical lifestyle in adulthood. It is therefore important that they develop physical literacy as well as a positive attitude towards physical activity. Unfortunately, despite its importance, physical literacy among university students is insufficiently investigated. In view of the above, this study employs a cluster randomized trial design to examine the effectiveness of sport education model delivered in the required physical education lessons at the university level to eligible students. The investigation focuses on the pre- and post-test and follow-up difference to see whether there are differences on perceived motivational climate, situational motivation, and their corresponding outcome of perceived PL, PA enjoyment and, self-report and objective PA levels. Also, this study investigates the fitness instruction time by videotaping and coding during every PE lesson from both groups. This study would be significant that the findings could establish the importance on physical literacy development through sport education model as well as develop students' physical literacy and positive attitude towards physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Physical education classes: universities in Hong Kong which are funded by the University Grants Committee and provides required PE lessons.
* Lecturers: graduated from master's degree or above, more than 5 years of teaching experience, in addition with the attendance of 12-hour continuing professional development workshop on Sport Education curriculum.
* Students: aged 18 or above, enrolled in 1-credit required physical education lessons and indicated all statements negatively in the self-screening Physical Activity Readiness Questionnaire (The Canadian Society for Exercise Physiology, 2017).

Exclusion Criteria:

* did not wish to participate;
* have currently used their own wearable activity tracker;
* indicated any major physical, psychiatric, or cardiovascular-related problems diagnosed by a physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Wai Raymond Sum, EdD, Principal Investigator — Chinese University of Hong Kong; Siu Ming Choi, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be provided after publication for 6 months.
Access Criteria: All IPD that underlie results in a publication will be available publicly.

REFERENCES:
- [Background] Booth M. Assessment of physical activity: an international perspective. Res Q Exerc Sport. 2000 Jun;71 Suppl 2:114-20. doi: 10.1080/02701367.2000.11082794. No abstract available. PMID 25680021
- [Background] Hastie, P., & Wallhead, T. (2015). Operationalizing physical literacy through sport education. Journal of Sport and Health Science, 4(2), 132-138. doi:10.1016/j.jshs.2015.04.001
- [Background] McKenzie, T. L., Sallis, J. F., & Nader, P. R. (1992). SOFIT: System for observing fitness instruction time. Journal of teaching in physical Education, 11(2), 195-205.
- [Background] Milton, D., Appleton, P. R., Bryant, A., & Duda, J. L. (2018). Initial Validation of the Teacher-Created Empowering and Disempowering Motivational Climate Questionnaire in Physical Education. Journal of Teaching in Physical Education, 37(4), 340-351.
- [Background] Motl RW, Dishman RK, Saunders R, Dowda M, Felton G, Pate RR. Measuring enjoyment of physical activity in adolescent girls. Am J Prev Med. 2001 Aug;21(2):110-7. doi: 10.1016/s0749-3797(01)00326-9. PMID 11457630
- [Background] Sum RK, Ha AS, Cheng CF, Chung PK, Yiu KT, Kuo CC, Yu CK, Wang FJ. Construction and Validation of a Perceived Physical Literacy Instrument for Physical Education Teachers. PLoS One. 2016 May 19;11(5):e0155610. doi: 10.1371/journal.pone.0155610. eCollection 2016. PMID 27195664
- [Background] Sum RKW, Cheng CF, Wallhead T, Kuo CC, Wang FJ, Choi SM. Perceived physical literacy instrument for adolescents: A further validation of PPLI. J Exerc Sci Fit. 2018 Apr;16(1):26-31. doi: 10.1016/j.jesf.2018.03.002. Epub 2018 Mar 14. PMID 30662489
- [Background] Whitehead, M. E. (2013). Stages in physical literacy journey. International Council of Sport Science and Physical Education Bulletin, 65, 51-55.
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Hallal PC, Andersen LB, Bull FC, Guthold R, Haskell W, Ekelund U; Lancet Physical Activity Series Working Group. Global physical activity levels: surveillance progress, pitfalls, and prospects. Lancet. 2012 Jul 21;380(9838):247-57. doi: 10.1016/S0140-6736(12)60646-1. PMID 22818937
- [Background] Ryan RM, Deci EL. Self-determination theory and the facilitation of intrinsic motivation, social development, and well-being. Am Psychol. 2000 Jan;55(1):68-78. doi: 10.1037//0003-066x.55.1.68. PMID 11392867
- [Background] Sum, K. W. R., Wallhead, T., Ha, S., & Sit, H. (2018). Effects of physical education continuing professional development on teachers' physical literacy and self-efficacy and students' learning outcomes. International Journal of Educational Research, 88, 1-8.

RESULTS

PARTICIPANT FLOW:
Groups:
- Sport Education Group: Each sport education season included ten 90-min lessons, 1-day per week with each season following the five-phase sequence of team selection, teacher-directed, preseason, formal competition, and a culminating event. Participants in each class were divided into teams for the duration of each season and assigned specific sport-related roles (e.g., coach, fitness trainer, equipment manager) at the end of the team selection phase. Students gradually increased their responsibility for learning and had equal opportunity to participate in every lesson with tasks progressing from drills to modified games and competitions to obtain more authentic sports experiences within the lessons. To evaluate model fidelity, a sample lesson from each phase of the sport education season was observed and coded by the primary researcher using the sport education benchmark observational instrument.
- Control Group: Participants within the control group classes attended PE classes where teachers used traditional teacher-directed methods to teach the specific activities. These lessons started with a teacher-directed warm-up routine, followed by direct instruction of skills practices, and games without a consistent team and modification to meet the objective of the courses. Within the direct teaching approach, the teacher was assigned responsibility for all task presentation components of the learning tasks. No student role responsibilities or student-directed tasks were included within this approach. Students within the intact class changed teams each lesson and scores were not formally recorded for the game outcomes.
Period: Overall Study
Arm/Group | Sport Education Group | Control Group
Started | 208 | 202
Post-intervention | 191 | 190
Completed | 188 | 184
Not Completed | 20 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sport Education Group | Control Group | Total
Number analyzed (Participants) | 188 | 184 | 372
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 188 | 184 | 372
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.53 (0.93) | 18.57 (1.04) | 18.55 (0.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 55 | 111
  Male | 132 | 129 | 261
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 182 | 174 | 356
  Non-Chinese | 6 | 10 | 16

OUTCOME MEASURES:

1. Primary Outcome: Self-report Physical Activity Levels
Description: The globally standardized and validated International Physical Activity Questionnaire - short form was used to measure self-reported physical activity levels. Four generic items of vigorous, moderate, walking and sitting were included to obtain the physical activity levels from the participants. Example items included: During the last 7 days, on how many days did you do vigorous physical activities like heavy lifting, digging, aerobics, or fast bicycling (vigorous)? They are required to answer the total duration of different types of physical activity which was at least 10 uninterrupted minutes in the last 7 days. The following values continue to be used for the analysis: Walking = 3.3 METs, Moderate PA = 4.0 METs and Vigorous PA = 8.0 METs. The metabolic equivalent minutes/ week (MET-minutes/week) was calculated by this formula: 8 * vigorous-intensity activity minutes * days + 4 * moderate-intensity activity minutes * days + 3.3 * walking-intensity activity minutes * days.
Time Frame: Change from Baseline Self-report Physical Activity Levels at the 10th lesson (11th week) and Follow-up at the 13th lesson (15th week)
Measure: Mean (Standard Deviation); unit: MET-minutes/week
Groups:
- Sport Education Group: Each sport education season included ten 90-min lessons, 1-day per week with each season following the five-phase sequence of team selection, teacher-directed, preseason, formal competition, and a culminating event (Hastie et al. 2014). Participants in each class were divided into teams for the duration of each season and assigned specific sport-related roles (e.g., coach, fitness trainer, equipment manager) at the end of the team selection phase. Students gradually increased their responsibility for learning and had equal opportunity to participate in every lesson with tasks progressing from drills to modified games and competitions to obtain more authentic sports experiences within the lessons. To evaluate model fidelity, a sample lesson from each phase of the sport education season was observed and coded by the primary researcher using the sport education benchmark observational instrument (Ko et al. 2006; Sinelnikov 2009).
Arm/Group | Sport Education Group | Control Group
Number analyzed (Participants) | 188 | 184
MET-minutes/week
  Baseline | 2114.83 (2201.86) | 2245.51 (2307.48)
  Post-intervention | 3334.41 (2473.12) | 3052.78 (2222.99)
  Follow-up | 3664.36 (2390.37) | 3016.31 (2354.32)

2. Primary Outcome: Objective Physical Activity Levels
Description: The accelerometers (Actigraph GT3X+) will be used in this study to measure the dynamic range from -6 to +6 with 3 axes and 3mg/ LSB of sensitivity. A sub-sample of 64 participants was randomly selected to wear accelerometers to measure their objective physical activity levels for at least 8 hours per day, in 7 consecutive days (ActiGraph LLC, Pensacola, FL, USA). The data will be uploaded onto the computer and analyzed by ActiLife 6 software. Only 47 of their data were analyzed because the participants met the eligibility of wearing at least 8 hours per day in at least 5 days. Participants' objective physical activity levels will be categorized as sedentary, light, moderate or vigorous. Accordingly, metabolic equivalents were calculated automatically in its software that a higher value represents a better outcome.
Time Frame: Change from Baseline Objective Physical Activity Levels at the 10th lesson (11th week) and Follow-up at the 13th lesson (15th week)
Measure: Mean (Standard Deviation); unit: Metabolic equivalents
Arm/Group | Sport Education Group | Control Group
Number analyzed (Participants) | 29 | 18
Metabolic equivalents
  Baseline | 1.32 (0.26) | 1.28 (0.14)
  Post-intervention | 1.34 (0.27) | 1.29 (0.14)
  Follow-up | 1.25 (0.28) | 1.19 (0.1)

3. Secondary Outcome: Motivational Climate
Description: The 34-item Empowering and Disempowering Motivational Climate Questionnaire in Physical Education was based on achievement goal theory and self-determination theory to assess students' perception of the motivational climate of empowering and disempowering features created by their physical education teachers. Participants responded to the instrument on a 1 to 5 Likert scale (1 = strongly disagree and 5 = strongly agree). The total subscale score range was 17 - 85 that higher values represent a better outcome in the empowering subscale and vice versa for the disempowering. Milton et al. (2018) clarified the questionnaire is internally consistent (α = 0.82 - 0.91) and factorial and construct validity. The empowering and disempowering scores were first summed up by their accordance item and the descriptive average scores were then calculated.
Time Frame: Baseline, 10th lesson (11th week) (Post-intervention) and 13th lesson (15th week) (Follow-up)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sport Education Group | Control Group
Number analyzed (Participants) | 188 | 184
score on a scale
  Empowering - Baseline | 62.97 (8.4) | 62.44 (9.08)
  Empowering - Post-intervention | 68.55 (8.14) | 67.48 (8.5)
  Empowering - Follow-up | 68.77 (8.53) | 67.45 (9.11)
  Disempowering - Baseline | 44.13 (10.74) | 41.95 (10.89)
  Disempowering - Post-intervention | 37.03 (10.64) | 37.96 (11.73)
  Disempowering - Follow-up | 37.18 (11.47) | 38.35 (11.12)

4. Secondary Outcome: Situational Motivation
Description: The Situational Motivation Scale was used to measure participants' situational intrinsic and extrinsic motivation while performing given physical activities. Participants responded to the instrument on a 7-point Likert scale (1 = not at all true and 7 = very true). The total subscale score range was 4 - 28 that higher values represent a better outcome for all subscales. Example items include: (a) this activity is fun (intrinsic motivation); (b) I believe this activity is important for me (identified regulation); (c) I don't have any choice (external regulation); and (d) I do this activity, but I am not sure it is a good thing to pursue it (amotivation). It illustrated that it has adequate internal consistency (α = 0.77-0.95) and construct validity in physical activity settings among college students aged from 18 - 22 years (mean age = 18.9). The motivational spectrum scores were first summed up by their accordance item and the descriptive average scores were then calculated.
Time Frame: Baseline, 10th lesson (11th week) (Post-intervention) and 13th lesson (15th week) (Follow-up)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sport Education Group | Control Group
Number analyzed (Participants) | 188 | 184
score on a scale
  Intrinsic motivation - Baseline | 19.82 (3.62) | 19.41 (3.86)
  Intrinsic motivation - Post-intervention | 20.98 (3.99) | 20.22 (4.28)
  Intrinsic motivation - Follow-up | 21.06 (3.85) | 20.57 (4.33)
  Identified regulation - Baseline | 19.59 (3.65) | 19.52 (3.76)
  Identified regulation - Post-intervention | 20.43 (4.04) | 19.96 (3.95)
  Identified regulation - Follow-up | 20.65 (3.93) | 20.34 (4.32)
  Extrinsic regulation - Baseline | 16.6 (4.22) | 17.14 (3.78)
  Extrinsic regulation - Post-intervention | 17.07 (3.78) | 17.73 (3.74)
  Extrinsic regulation - Follow-up | 17.24 (4.14) | 17.96 (3.7)
  Amotivation - Baseline | 12.88 (4.4) | 13.37 (4.61)
  Amotivation - Post-intervention | 12.83 (4.79) | 13.32 (4.72)
  Amotivation - Follow-up | 12.6 (4.71) | 13.24 (5.16)

5. Secondary Outcome: Perceived Physical Literacy
Description: The Perceived Physical Literacy Instrument is a 9-item instrument which is used to measure both teachers' and adolescents' perceived physical literacy. Participants responded to the instrument on a 1 to 5 Likert scale (1 = strongly disagree and 5 = strongly agree). The total subscale score range was 3 - 15 that higher values represent a better outcome for all subscales. Example statements include: (a) I am physically fit, in accordance with my age (sense of self and self-confidence); (b) I have strong social skills (self-expression and communication with others); (c) I am aware of the benefits of sports related to health (knowledge and understanding). The scale scores are reliable with the internal consistency from .73 to .76. The scores were first summed up by their accordance item and the descriptive average scores were then calculated.
Time Frame: Baseline, 10th lesson (11th week) (Post-intervention) and 13th lesson (15th week) (Follow-up)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sport Education Group | Control Group
Number analyzed (Participants) | 188 | 184
score on a scale
  Sense of self and self-confidence - Baseline | 9.52 (2.44) | 9.57 (2.48)
  Sense of self and self-confidence - Post-intervention | 9.85 (2.41) | 9.64 (2.5)
  Sense of self and self-confidence - Follow-up | 9.92 (2.45) | 10.04 (2.51)
  Self-expression and communication with others - Baseline | 9.52 (2.29) | 9.5 (2.21)
  Self-expression and communication with others - Post-intervention | 9.87 (2.4) | 9.62 (2.19)
  Self-expression and communication with others - Follow-up | 10.04 (2.4) | 9.77 (2.3)
  Knowledge and understanding - Baseline | 11.11 (2.11) | 1122 (2.11)
  Knowledge and understanding - Post-intervention | 11.29 (2.1) | 11.05 (2.21)
  Knowledge and understanding - Follow-up | 11.28 (2.12) | 11.37 (2.2)

6. Secondary Outcome: Physical Activity Enjoyment
Description: The Physical Activity Enjoyment Scale is designed to measure how much a student enjoys participating in physical activity. Participants responded to the 16-items instrument on a 5-point Likert scale (1 = disagree a lot and 5 = agree a lot). The total subscale score range was 9 - 45 for positive and 7 - 35 for negative that higher values represent a better outcome in the positive subscale and vice versa for the negative. There are nine positive items such as "I find it pleasurable", "It gives me energy" and seven negative items such as "I dislike it", "It is not fun at all". Participants receive high scores on positive items and low scores on negative items would indicate a high enjoyment of physical activity. Motl et al. (2001) established adequate internal consistency (α = 0.81-0.86), and factorial and construct validity. The positive and negative scores were first summed up by their accordance item and the descriptive average scores were then calculated.
Time Frame: Baseline, 10th lesson (11th week) (Post-intervention) and 13th lesson (15th week) (Follow-up)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sport Education Group | Control Group
Number analyzed (Participants) | 188 | 184
score on a scale
  Positive - Baseline | 33.11 (5.96) | 32.46 (5.82)
  Positive - Post-intervention | 34.34 (6.04) | 33.58 (5.89)
  Positive - Follow-up | 34.44 (5.87) | 33.68 (6.25)
  Negative - Baseline | 14.55 (4.31) | 15.22 (4.47)
  Negative - Post-intervention | 14.09 (4.62) | 15.06 (4.67)
  Negative - Follow-up | 14.29 (4.81) | 15.14 (4.65)

7. Secondary Outcome: Fitness Instruction Time of Physical Education Lessons
Description: The Fitness instruction time was measured using the System for Observing Fitness Instruction Time (SOFIT; McKenzie et al., 1992) which is a validated and reliable momentary time sampling and interval observation instrument to gather quantitative data for assessing physical activity during PE lessons. SOFIT includes three intensities of students' physical activity levels, lesson context, and teacher behavior. Each category is coded using interval coding every 20 seconds (10 seconds observe; 10 seconds record) throughout the lesson. The observer decides on what is occurring at the moment an observation interval ends. Physical activity level, lesson content, and teacher behavior were measured as a percentage of physical education lesson time. Each outcome measure was then measured by averaging the percentage of physical education lesson time across the first to the tenth lesson.
Time Frame: The 1st lesson (Baseline) to the 10th lesson (11th week)
Measure: Mean (Standard Deviation); unit: percentage of lesson time
Arm/Group | Sport Education Group | Control Group
Number analyzed (Participants) | 188 | 184
percentage of lesson time
  PA levels - Lying down | 0.11 (0.47) | 0.11 (0.35)
  PA levels - Sitting | 12.35 (11.46) | 12.78 (10.83)
  PA levels - Standing | 48.77 (23.28) | 47.54 (20.99)
  PA levels - Walking | 27.32 (11.44) | 29.13 (10.64)
  PA levels - Vigorous | 11.45 (13.25) | 10.45 (10.96)
  Lesson context - General content | 18.62 (8.8) | 14.17 (5.45)
  Lesson context - Knowledge content | 16.93 (10.62) | 24.01 (8.97)
  Lesson context - Fitness | 7.27 (10.91) | 5.26 (4)
  Lesson context - Skill practice | 34.37 (15.79) | 37.36 (13.91)
  Lesson context - Game play | 19.1 (14.6) | 16.09 (12.79)
  Lesson context - Other | 3.71 (11.29) | 3.07 (10.99)
  Teacher behavior - Promotes fitness | 0.56 (1.2) | 0.61 (1.2)
  Teacher behavior - Demonstrates fitness | 1.99 (9.84) | 1.63 (3.4)
  Teacher behavior - Instructs generally | 38.57 (15.9) | 47.53 (15.92)
  Teacher behavior - Manages | 26.3 (12.21) | 22.26 (14.41)
  Teacher behavior - Observes | 31.71 (14.18) | 27.07 (14.87)
  Teacher behavior - Other task | 0.87 (1.76) | 0.09 (2.04)

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious, and other adverse events were not collected.
Description: All-cause mortality, serious, and other adverse events were not collected.
Arm/Group | Sport Education Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-09-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT03888885/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT03888885/SAP_001.pdf
  • Informed Consent Form (2021-09-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT03888885/ICF_002.pdf